CLINICAL TRIAL: NCT07287813
Title: Pharmacokinetics/Pharmacodynamics and Therapeutic Drug Monitoring of Novel β-lactams and β-lactamase Inhibitors in Critically Ill Patients Undergoing Extracorporeal Therapy
Brief Title: Extracorporeal Therapy and Therapeutic Drug Monitoring
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Simona De Gregori, PhD in Chemical Sciences, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: BL/BLIs in ICU - 2024
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-08

CONDITIONS: ICU Patients With ECMO And-or RRT and With Gram Negative Infections Susceptible to BL-BLIs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to comparatively evaluate serum concentrations of continuously applied antibiotics in ICU patients, with and without ECMO/RRT support.

DETAILED DESCRIPTION:
Among all patients being treated with new generation antibiotics (beta.lactams and beta-lactamase inhibitors), we will take into consideration the results of those admitted to intensive care units.

Effective antimicrobial treatment is critical to reduce their mortality associated with bacterial sepsis. They often also require extracorporeal supports, such as renal replacement therapy (RRT) and extracorporeal membrane oxygenation (ECMO), for their survival. However, few studies, limited only to some drugs, report the importance of therapeutic drug monitoring for adequate dose adjustment in these particular conditions of extracoporeal support.

The risk of reaching sub therapeutic or toxic levels is quite high, due to possible very significant variations in the pharmacokinetics of the drugs because of their interaction with the various components of the ECMO and RRT devices, the characteristics of the drug itself and the pathophysiological changes of the patients on ECMO and/or RRT.

Primary aim is to evaluate whether the standard prescriptions of beta lactams/beta lactamase inhibitors (BL/BLIs) are adequate to achieve the optimal PK/PD target also for ECMO and RRT (or combined) patients admitted to intensive care unit.

Secondary aims include to evaluate:

* the occurrence of sub-therapeutic and/or toxic drugs levels
* the proportion of patients with insufficient drugs levels in different subgroups (i.e., absence of extracorporeal therapy vs. ECMO; absence of extracorporeal therapy vs. RRT, absence of extracorporeal therapy vs ECMO and RRT) - the proportion of patients with toxic or sub-therapeutic drugs levels in the same subgroups;
* the proportion, when possible, of drugs level before and during the extracorporeal therapy, for the same patient;
* the occurrence of drug resistance by pathogens and their mechanism

ELIGIBILITY:
Inclusion Criteria:

* adult patients (age 18y or older)
* admitted to ICU
* supported or not-supported with extracorporeal membrane oxygenation (ECMO) and/or renal replacement therapy (RRT)
* affected by gram-negative bacterial infections susceptible to the novel antibiotics.

Exclusion Criteria:

* Pediatric age (<18y)
* allergies to pharmaceutical and/or inactive drug ingredients (excipients)
* life expectancy less than 1 month
* body mass index (BMI) >45 kg/m2
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients with ECMO and/or RRT and with gram-negative infections susceptible to BL/BLIs
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-12-12 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Primary aim | up to 24 months
  evaluate whether the standard prescriptions of beta lactams/beta lactamase inhibitors (BL/BLIs) are adequate to achieve the optimal PK/PD target also for ECMO and RRT (or combined) patients admitted to intensive care unit.

SECONDARY OUTCOMES:
occurrence of sub-therapeutic and/or toxic drugs levels | up to 24 months
proportion of patients with insufficient drugs levels in different subgroups | up to 24 months
proportion of patients with toxic or sub-therapeutic drugs levels in the same subgroups | up to 24 months
proportion, when possible, of drugs level before and during the extracorporeal therapy, for the same patient | up to 24 months
occurrence of drug resistance by pathogens and their mechanism | up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy, Italy